CLINICAL TRIAL: NCT00585546
Title: Harefield Recovery Protocol Study (HARPS): A Nonrandomized, Open Label, Multicenter Evaluation of Potential Recovery of Heart Function in Patients With Refractory Chronic Heart Failure by Treatment With Combination of Left Ventricular Assist Device (LVAD), Drugs to Induce Maximal Reverse Remodeling and the Beta-2 Adrenergic Receptor Agonist Clenbuterol.
Brief Title: Harefield Recovery Protocol Study for Patients With Refractory Chronic Heart Failure
Acronym: HARPS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No longer could obtain clenbuterol
Sponsor: Francis D. Pagani (Other)
Collaborators: Georgetown University (Other); Montefiore Medical Center (Other); Northwestern University (Other); Ohio State University (Other); Texas Heart Institute (Other); University of Minnesota (Other); University of Pennsylvania (Other); Thoratec Corporation (Industry)
Responsible Party: Sponsor-Investigator, Francis D. Pagani, Professor of Cardiac Surgery, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HARPS; NCT00701116 (obsolete NCT alias)
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Heart Failure; Dilated Cardiomyopathy
Keywords: heart failure; dilated cardiomyopathy; heart assist device; clenbuterol; adrenergic beta agonists; heart transplantation
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated | interventions — Clenbuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LVAD and Clenbuterol (Experimental)
  Interventions: Drug: clenbuterol

INTERVENTIONS:
Drug: clenbuterol — Clenbuterol 20 mcg tablets uptitrated from 20 mcg PO TID to a maximally tolerated dose not to exceed 700 mcg PO TID. Patients will then be switched to the equivalent dose of clenbuterol liquid 59 mcg/ml PO TID. Clenbuterol will be administered for a minimum of 3 months and a maximum of 12 months.
  Other Names: Spiropent

SUMMARY:
The purpose of this study is to evaluate whether patients with chronic heart failure not due to coronary artery disease who require use of a left ventricular assist device (LVAD) for refractory heart failure can recover sufficient heart function to allow the pump to be explanted. The study aims to avoid the need for transplantation in these patients by using standard heart failure medications to reduce the size of the left ventricle and then using the investigational drug, clenbuterol, to further improve left ventricular function.

DETAILED DESCRIPTION:
The hypothesis of this study is that patients with dilated nonischemic cardiomyopathy who require support with an implanted left ventricular assist device (LVAD) for chronic refractory heart failure can, with a specific two-staged medical regimen designed to enhance maximal reverse remodeling (an angiotensin converting enzyme inhibitor, beta blocker, angiotensin receptor blocker, aldosterone antagonist and digoxin [stage 1]) and prevent/reverse myocardial atrophy (the β2 agonist clenbuterol [stage 2]), recover adequate left ventricular systolic function to allow LVAD explantation and subsequent intermediate-term survival without need for mechanical circulatory support or heart transplantation.

Within one year of this study's start, a new LVAD became the standard of care for implantation, so the study device became an inferior standard of care shortly thereafter. By 2012 the trial was stopped for futility in enrollment. Thus, certain original outcomes have been deleted, specifically because there was only a single subject explanted, multivariate analysis for sustainability of reverse remodeling following LVAD explantation and predictors of recovery of left ventricular function/remodeling and of LVAD removal could not be done.

Similarly, and for lack of funding, biobank components were not collected; therefore no data exists to present biochemical, structural, cellular and molecular changes in the myocardium resulting from the HARPS protocol interventions, changes in systemic inflammation, circulating progenitor cells and growth factors, or DEXA scan based data: changes in body mass, lean muscle mass, muscle strength and maximal and submaximal exercise capacity. All remaining outcome measures have been edited to more precisely show the outcome measures intended.

ELIGIBILITY:
Inclusion Criteria:

Patients with refractory symptomatic heart failure (NYHA Class IV, or Stage D) due to dilated, non-ischemic cardiomyopathy who meet the following criteria:

* Severe clinical heart failure with associated haemodynamic compromise resistant to intensive medical therapy and requiring LVAD implantation
* Duration of heart failure symptoms to be ≥ 12 months prior to LVAD implant
* Documentation of LVEF ≤ 40% at least 1 year prior to LVAD implantation
* LVEF ≤ 30% and cardiomegaly at the time of LVAD implantation as documented by radionuclide or contrast ventriculography or by echocardiography
* Nonischemic etiology confirmed by coronary angiography within two years of enrollment
* Listed for heart transplantation or plan to list for heart transplantation pending successful LVAD implantation in one of the participating centers, as per usual transplant listing policy at each participating center
* >= 18 years of age
* Body surface area >= 1.5 m2
* Have an implantable defibrillator in place or a commitment to implant an ICD prior to hospital discharge
* Have undergone insertion within prior 2 weeks or will be inserted with a Heartmate XVE LVAD with use of antimicrobial prophylaxis and drive line restraining belt

Exclusion Criteria:

* Not a heart transplant candidate
* Evidence of active acute myocarditis
* Pulmonary Vascular Resistance > 6 Wood Units
* History of previous CVA resulting in significant fixed motor deficit limiting ability to perform exercise testing
* Previous prosthetic replacement of aortic and/or mitral valve(s)
* Hypertrophic obstructive cardiomyopathy
* LVIDD < 5 cm by surface echocardiogram (restrictive cardiomyopathy)
* Irreversible multi-organ failure
* Underlying bleeding disorder, or platelet count < 75,000, INR > 2.5 (without Coumadin), or Hgb < 8.0.
* Pregnant or lactating women or unwilling to utilize two reliable methods of birth control for women of childbearing age
* Receipt of other investigational drug therapy during LVAD support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie W. Miller, MD, Principal Investigator — Georgetown University; Keith D. Aaronson, MD, MS, Study Director — University of Michigan; Francis D. Pagani, MD, PhD, Study Director — University of Michigan
Locations (7):
- United States (7):
  - Georgetown Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Birks EJ, Tansley PD, Hardy J, George RS, Bowles CT, Burke M, Banner NR, Khaghani A, Yacoub MH. Left ventricular assist device and drug therapy for the reversal of heart failure. N Engl J Med. 2006 Nov 2;355(18):1873-84. doi: 10.1056/NEJMoa053063. PMID 17079761

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 19 consented, 1 was a screen fail and did not enter the study protocol.
Groups:
- LVAD and (Intended) Clenbuterol: Participants, all of whom received LVAD implantation, were to begin clenbuterol treatment 12 weeks after their implantation.
  Clenbuterol 20 mcg tablets uptitrated from 20 mcg PO TID to a maximally tolerated dose not to exceed 700 mcg PO TID. Patients will then be switched to the equivalent dose of clenbuterol liquid 59 mcg/ml PO TID. Clenbuterol will be administered for a minimum of 3 months and a maximum of 12 months.
Period: LVAD Implantation Required for 4 Months
Arm/Group | LVAD and (Intended) Clenbuterol
Started | 18
Completed | 13
Not Completed | 5
Period: Clenbuterol Treatment - up to 12 Months
Arm/Group | LVAD and (Intended) Clenbuterol
Started | 13
Completed | 9
Not Completed | 4
Not completed — Death | 1
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [54 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects Who Experience LVAD Removal and Subsequent Freedom From Mechanical Circulatory Support or Heart Transplantation for 1-year After Explantation
Time Frame: One year after LVAD explant or until transplant or death (if not explanted)
Measure: Number; unit: percentage of participants
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 18
percentage of participants | 5.6

2. Secondary Outcome: The Number of Evaluable Subjects Meeting Explant Criteria and Subsequently Explanted
Time Frame: Maximum 12 months after LVAD implantation
Population: Because only 13 began Clenbuterol, only 13 are "evaluable" for this purpose.
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 13
Participants | 1

3. Secondary Outcome: Number of Subjects Who Received Maximum Target Dose of Clenbuterol
Time Frame: Up to 16 months after LVAD implantation (12 months after beginning clenbuterol)
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 13
Participants | 13

4. Secondary Outcome: Time to Device Explant for Subjects Meeting Explant Criteria Defined in the Protocol
Description: Time from LVAD placement to explant for the single participant who achieved explant
Time Frame: Time to explant (but not to be followed for more than 16 months)
Measure: Number; unit: weeks
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 1
weeks | 28

5. Secondary Outcome: Absolute Change in Left Ventricular Ejection Fraction From Explant to 18 Months Following Device Explant
Time Frame: 18 months after explantation
Measure: Number; unit: absolute change in ejection fraction
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 1
absolute change in ejection fraction | -.09

6. Secondary Outcome: Absolute Percent Change in Serum Creatinine and Aspartate Transaminase (AST) From Baseline to Week 8 Post Implant
Time Frame: Up to 8 weeks after LVAD implantation
Population: Because data only is available for 15 participants for 8 week post implant AST value, it has a different participants analyzed value
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 18
percent change
  Creatinine | 17.2 (15.2)
  aspartate transaminase (AST): number analyzed (Participants) | 15
  aspartate transaminase (AST) | 25 (19.7)

7. Secondary Outcome: Mean Change in EuroQoL Visual Analog Scale (EQ5D-VAS) From Baseline to 6 Months and 1 Year Following Device Implant
Description: Scale 0 - 100 where 0 is worst possible health state and 100 is perfect health.
Time Frame: 1 year following LVAD implantation
Population: While baseline data was available for 13 participants at baseline, (start of clenbuterol), different numbers of participants provided evaluable data At six months post implant and 12 months, so the mean changes are based on the actual population that provided both data points as listed below
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 13
units on a scale
  6 months post implant: number analyzed (Participants) | 7
  6 months post implant | 46 (35)
  12 months post implant: number analyzed (Participants) | 12
  12 months post implant | 51 (30)

8. Secondary Outcome: Mean Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) From Baseline to 6 Months
Description: Scale 0 - 105 (0- 5 on 21 items) where 0 means heart failure has not limited daily life at all and high scores mean that daily functions are greatly limited.
Time Frame: 6 months following LVAD implantation
Population: Only 11 participants provided usable data at the six month time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 11
units on a scale | 28.3 (19.7)

9. Secondary Outcome: Mean Change in Left Ventricular Ejection Fraction From Device Implant to Completion of Clenbuterol Therapy
Time Frame: up to 16 months, variable based on length of time receiveing clenbuterol
Population: data is available for 9 evaluable subjects at end of clenbuterol
Measure: Mean (Standard Deviation); unit: ejection fraction
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 9
ejection fraction | 0.16 (.10)

10. Secondary Outcome: Absolute Percent Change in Serum Creatinine and Aspartate Transaminase (AST) From Baseline to Week 8 Post Clenbuterol
Time Frame: baseline to week 8 post clenbuterol
Population: baseline data is based on 19 participants, but different subsequent data collections had different numbers of evaluable subjects listed below
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 19
percent change
  creatinine from baseline to week 8 of clenbuterol: number analyzed (Participants) | 10
  creatinine from baseline to week 8 of clenbuterol | -15.8 (13.3)
  AST from baseline to week 8 on clenbuterol: number analyzed (Participants) | 9
  AST from baseline to week 8 on clenbuterol | 15.6 (14.3)

11. Secondary Outcome: Mean Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) From Baseline to 1 Year Following Device Implant
Description: as for outcome 8
Time Frame: 1 year
Population: Data is not available for Minnesota Living with Heart Failure Questionnaire at the 12 month time point.
Arm/Group | LVAD and Clenbuterol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for approximately 24 months or up to transplant, death, or explant
Arm/Group | LVAD and Clenbuterol
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 13/18
Other Adverse Events (participants affected / at risk) | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LVAD and Clenbuterol (N=18)
Abdominal Perforation Requiring Re-Operation (Gastrointestinal disorders) | 1
Anemia, Pancytopenia (Blood and lymphatic system disorders) | 1
AV Endocarditis (Infections and infestations) | 1
Bleeding (Gastrointestinal disorders) | 4
Cardiac arrhythmia (Cardiac disorders) | 2
Cardiopulmonary Arrest (Cardiac disorders) | 1
Dehydration (Renal and urinary disorders) | 1
Device malfunction (Product Issues) | 2
Fever (Infections and infestations) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
History Afib/Flutter since XVE Implant (Cardiac disorders) | 1
Infection (Infections and infestations) | 3
Intermittent Fever, Pain, Leukocytosis (Infections and infestations) | 1
Left Atrial Thrombus (Cardiac disorders) | 1
Left Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Left Sided Pain Radiating to Axilla (Injury, poisoning and procedural complications) | 1
Left sided pneumothorax - Left Pleural CT inserted (Injury, poisoning and procedural complications) | 1
Nausea and Vomiting (Gastrointestinal disorders) | 1
Neurological event (Nervous system disorders) | 3
Renal dysfunction (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Retropericardial Hematoma (Injury, poisoning and procedural complications) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Viral Syndrome (Infections and infestations) | 1
Pericardial fluid collection (Cardiac disorders) | 1
Heart Failure (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LVAD and Clenbuterol (N=18)
Abdominal Pain (Gastrointestinal disorders) | 1
Bleeding (Gastrointestinal disorders) | 1
Cardiac arrhythmia (Cardiac disorders) | 1
Chest Pain (Cardiac disorders) | 1
Elevated White Blood Cell/Leukocytosis (Infections and infestations) | 1
Hyperkalemia (Renal and urinary disorders) | 1
Hypertension (Cardiac disorders) | 2
Implantable Cardioverter Defibrillator (ICD) Discharge (Cardiac disorders) | 1
Infection (Infections and infestations) | 4
Muscle Pain (Injury, poisoning and procedural complications) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neurological (Nervous system disorders) | 2
Psychiatric episode (Psychiatric disorders) | 1
Severe Muscle Spasms (Injury, poisoning and procedural complications) | 1
Sinus Tachycardia Leading to ICD Shocks (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Blood Bowel Movement (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Because a new standard of care was developed during the start of the trial, the trial was stopped for futility in enrollment. The public should exercise great caution in drawing conclusions from such a small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes